CLINICAL TRIAL: NCT06598436
Title: Achieving Chronic Care equiTy by leVeraging the Telehealth Ecosystem
Acronym: ACCTiVATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Tech Council (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-40207; R01MD019042 (NIH)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Diabetes
Keywords: Adverse Event; Blood Pressure; Community Advisory Board (CAB); Chronic Kidney Disease (CKD); Clinic-level Intervention; Clinical Research Coordinator (CRC); Cardiovascular Disease; Digital Coach Navigator; Federally Qualified Health Center (FQHC); Good Clinical Practice; Health Care Systems; Health Insurance Portability and Accountability Act of 1996; Hemoglobin A1C; Informed Consent Form (ICF); Institutional Review Board (IRB); Library; National Institutes of Health (NIH); Randomized Control Trial (RCT); National Institute of Minority Health and Health Disparities (NIHMD); Patient Advisory Council (PAC); Patient-level Intervention; Principal Investigator (PI); Socioeconomic Status; San Francisco Health Network (SFHN); Systolic Blood Pressure (SBP); Telehealth; Telemedicine; University of California, San Francisco (UCSF); Zuckerberg San Francisco General Hospital (ZSFG)
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The investigators propose a prospective, multilevel, nonblinded 2x2 randomized controlled trial to determine the effectiveness of a clinic-level intervention and a patient-level intervention, as well as the potential synergistic impact of both interventions on process outcomes and clinical measures of diabetes control. Five of the 11 participating clinics will be randomized to receive practice facilitation for 24 months. After implementing the clinic-level intervention, the investigators will begin recruiting/randomizing eligible patients in a 1:2 ratio to receive tailored digital coaching (n=200) or usual care (n=400) for 3 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient Intervention + Clinic Intervention (Experimental): Digital coach navigator + Clinic Intervention
  Interventions: Other: Digital Health Coaching (Patient-Level Intervention); Other: Practice Facilitation (Clinic-Level Intervention)
- Patient Usual Care + Clinic Usual Care (No Intervention): Usual Care (Patient-Level) + Clinic Usual Care
- Patient Intervention + Clinic Usual Care (Experimental): Digital coach navigator + Clinic Usual Care
  Interventions: Other: Digital Health Coaching (Patient-Level Intervention)
- Patient Usual Care + Clinic Intervention (Experimental): Usual Care (Patient-Level) + Clinic Intervention
  Interventions: Other: Practice Facilitation (Clinic-Level Intervention)

INTERVENTIONS:
Other: Digital Health Coaching (Patient-Level Intervention) — The patient-level intervention combines the role of digital health navigator and chronic disease health coach to facilitate access to devices and broadband, offer digital skills training, and provide chronic disease health coaching focused on telehealth modalities.
  Arms: Patient Intervention + Clinic Intervention; Patient Intervention + Clinic Usual Care
Other: Practice Facilitation (Clinic-Level Intervention) — The clinic-level intervention includes primary care clinic support through practice facilitation that empowers team members to address racial/ethnic disparities in telehealth use through consistent review of telehealth equity data and input from clinic-specific Patient Advisory Councils (PACs).
  Arms: Patient Intervention + Clinic Intervention; Patient Usual Care + Clinic Intervention

SUMMARY:
This study examines the impact of a multi-level intervention aiming to improve telehealth access for low-income patients managing chronic health conditions, such as hypertension and diabetes. The multi-level intervention includes clinic-level practice facilitation and patient-level digital health coaching.

DETAILED DESCRIPTION:
ACCTIVATE is a multi-level intervention (including practice facilitation and patient digital coaching) that aims to tackle patient-level and clinic-level barriers to increase the equitable use of telehealth tools for chronic disease management. Direct patient support via digital coaching can meet the needs of patients who have been left behind in the digital divide. For those with reduced digital literacy and low access to smartphones and broadband, this resource can increase their confidence in using digital technologies and engaging in virtual care. Additionally, primary care clinic support through practice facilitation can empower team members to address racial/ethnic disparities in telehealth use through equitable screening/offering of digital technologies, resources to prepare patients for virtual chronic disease management, and consistent review of telehealth equity data. The investigators hypothesize that this multi-level intervention will improve patient control of chronic health conditions (i.e., glycosylated hemoglobin) as well as digital literacy, while also increasing patient and clinician engagement with patient portals, telehealth video visits and remote monitoring.

Aim 1: Assess the impact of the multi-level intervention on clinical outcomes at 3, 6, 12, and 24 months. Our working hypotheses are that patients randomized to receive digital coaching (vs. usual care) will experience a greater change in mean glycosylated hemoglobin A1C, both overall and among Black and Latinx patients. Clinics randomized to practice facilitation (vs. usual care) will experience a greater clinic-level change in mean glycosylated hemoglobin A1C, both overall and among their Black and Latinx populations.

Aim 2: Assess the impact of the multi-level intervention on process outcomes related to digital literacy, engagement in care, and health IT utilization at 3, 6, 12, and 24 months. The investigators hypothesize that randomization to digital coaching (vs. usual care) will increase patient portal use, digital literacy, and visit show rate, overall and among Black and Latinx patients. Randomization to practice facilitation (vs. usual care) will increase clinic-level use of telehealth video visits and patient-portal communication, overall and with Black and Latinx patients.

Aim 3: Conduct a mixed methods evaluation of intervention implementation outcomes. Quantitative engagement data, direct observations of intervention sessions, and stakeholder interviews will characterize implementation outcomes and factors necessary to integrate the multi-level intervention into clinical operations, applying the RE-AIM implementation science framework.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* English or Spanish-Speaking
* Have uncontrolled diabetes defined as a listed diagnosis of diabetes with a recorded A1C ≥ 8.0% in the past two years or have uncontrolled HTN defined as a listed diagnosis of HTN and last recorded documented SBP >140 mmHg
* At least 2 visits at a participating SFHN primary care site in the last 24 months

Exclusion Criteria:

* Higher than average digital literacy, defined as an Digital Healthcare Literacy Scale (DHLS) score greater than 10, as determined prior to the baseline study visit; these patients may not benefit from a digital coaching intervention.
* Presence of co-morbid conditions that would make it inappropriate to focus on telehealth chronic disease management. Conditions may include: end-stage or terminal condition with limited life expectancy and severe mental illness.
* Lack of any working phone number
* Visual or hearing impairment that precludes use of telehealth for chronic disease management
* Cognitive impairment defined by the inability to restate study goals during the consent process
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Level Hemoglobin A1C | Baseline, month 3, month 6, and month 12
  Change in A1C (%) will be determined by subtracting month 3, 6, and 12 A1C values from baseline A1C
Change in Patient Portal Use | Baseline, month 3, month 6, and month 12
  The average number of patient portal log-ins per month will be obtained from the EHR

SECONDARY OUTCOMES:
Digital Literacy | Baseline, month 3, month 6, and month 12
  Digital literacy will be ascertained with the Digital Healthcare Literacy Scale (DHLS). The DHLS is an 3-item scale that uses a 5-point Likert scale. Scores range from 0 to 12, with higher scores indicating higher digital health care literacy.
  Ongoing digital literacy will be ascertained with the Digital Equity Screening Tool Scale (DEST). The DEST is an 5-item scale that uses a 5-point Likert scale.
Medication Adherence | Baseline, month 3, month 6, and month 12
  Medication adherence will be ascertained by the eight-item Morisky Medication Adherence Scale (MMAS-8). The scales score ranges from 0 to 8, with higher scores indicating greater medication adherence.
  High adherence: A score of 8 Medium adherence: A score of 6-8 Low adherence: A score of 6 and below.
Patient Activation Measure (PAM) | Baseline, month 3, month 6, and month 12
  Patient activation will be measured by the Patient Activation Measure (PAM). The PAM-13 consists of 13 items on a 4-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree, 0 = undecided). Item scores are summed to a raw score resulting in theoretical values between 13 and 52, with higher scores indicating higher patient activation.
Change in Clinic-Wide Blood Pressure (mmHg) | Baseline, month 3, month 6, month 12, and month 24
  BP readings will be obtained from the EHR
Change in Clinic-Wide Hemoglobin A1C (average) | Baseline, month 3, month 6, month 12, and month 24
  Hemoglobin A1C readings will be obtained from the EHR
Change in Patient-Level Systolic BP (mmHg) | Baseline, month 3, month 6, month 12
  Changes in mean SBP from baseline, using values from the electronic health record.
Proportion of Primary care Clinic Visits Completed by Video | Baseline, month 3, month 6, month 12 and month 24
  This proportion will be ascertained from the electronic health record.
Number of Patient Portal Communications Completed by Primary Care Team Members | Baseline, month 3, month 6, month 12, and month 24
  The number of patient portal communications will be ascertained from the EHR
Clinic-level Visit Show Rates | Baseline, month 3, month 6, month 12, and month 24
  Visit show rates for in-person, phone, or telehealth video as obtained from the EHR
Change in Patient-Level urine microalbuminuria (mg/g) among individuals with hypertension and/or diabetes | Baseline, month 3, month 6, month 12
  Urine microalbuminuria (mg/g) will be obtained from the electronic health record.
Change in Clinic-Wide Urine Albumin-Creatinine Ratio UACR (mg/g) among individuals with hypertension and/or diabetes. | Baseline, month 3, month 6, month 12, and month 24
  Microalbuminuria values among individuals with hypertension and/or diabetes will be obtained from the EHR.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Tuot, MD MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital (ZSFG) & SF Department of Public Health (DPH), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from approximately 690 participants recruited from primary care clinics in the San Francisco Health Network with uncontrolled diabetes (defined as glycosylated A1c greater than or equal to 8.0%). The final dataset will include self-reported demographic, telehealth engagement, and chronic disease self-management data from self-report, and additional demographic, clinical outcome, and telehealth utilization data from the electronic medical record. The data will be made available in a de-identified format in a .csv or .dta file. In addition to the IPD data set, the ACCTIVATE study team will share the data set, data dictionary, statistical analysis plan, analytic code, and final protocol with amendments
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available as soon as possible or at the time of associated publication. The duration of preservation and sharing of the data will be a minimum of 5 years after the end of the funding period.
Access Criteria: The investigators plan to provide access to the data via Dryad. Anyone can download a dataset via Dryad in the form of a zip file. Dryad will maintain storage and access of the data for as long as it maintains scientific utility.

REFERENCES:
- [Background] Patrick K, Norman GJ, Davila EP, Calfas KJ, Raab F, Gottschalk M, Sallis JF, Godbole S, Covin JR. Outcomes of a 12-month technology-based intervention to promote weight loss in adolescents at risk for type 2 diabetes. J Diabetes Sci Technol. 2013 May 1;7(3):759-70. doi: 10.1177/193229681300700322. PMID 23759410
- [Background] Grossman LV, Masterson Creber RM, Benda NC, Wright D, Vawdrey DK, Ancker JS. Interventions to increase patient portal use in vulnerable populations: a systematic review. J Am Med Inform Assoc. 2019 Aug 1;26(8-9):855-870. doi: 10.1093/jamia/ocz023. PMID 30958532
- [Background] Irizarry T, Shoemake J, Nilsen ML, Czaja S, Beach S, DeVito Dabbs A. Patient Portals as a Tool for Health Care Engagement: A Mixed-Method Study of Older Adults With Varying Levels of Health Literacy and Prior Patient Portal Use. J Med Internet Res. 2017 Mar 30;19(3):e99. doi: 10.2196/jmir.7099. PMID 28360022
- [Background] Taha J, Sharit J, Czaja SJ. The impact of numeracy ability and technology skills on older adults' performance of health management tasks using a patient portal. J Appl Gerontol. 2014 Jun;33(4):416-36. doi: 10.1177/0733464812447283. Epub 2012 Jun 4. PMID 24781964
- [Background] Sarkar U, Karter AJ, Liu JY, Adler NE, Nguyen R, Lopez A, Schillinger D. Social disparities in internet patient portal use in diabetes: evidence that the digital divide extends beyond access. J Am Med Inform Assoc. 2011 May 1;18(3):318-21. doi: 10.1136/jamia.2010.006015. Epub 2011 Jan 24. PMID 21262921
- [Background] Wallace LS, Angier H, Huguet N, Gaudino JA, Krist A, Dearing M, Killerby M, Marino M, DeVoe JE. Patterns of Electronic Portal Use among Vulnerable Patients in a Nationwide Practice-based Research Network: From the OCHIN Practice-based Research Network (PBRN). J Am Board Fam Med. 2016 Sep-Oct;29(5):592-603. doi: 10.3122/jabfm.2016.05.160046. PMID 27613792
- [Background] Sarkar U, Karter AJ, Liu JY, Adler NE, Nguyen R, Lopez A, Schillinger D. The literacy divide: health literacy and the use of an internet-based patient portal in an integrated health system-results from the diabetes study of northern California (DISTANCE). J Health Commun. 2010;15 Suppl 2(Suppl 2):183-96. doi: 10.1080/10810730.2010.499988. PMID 20845203
- [Background] Lyles CR, Tieu L, Sarkar U, Kiyoi S, Sadasivaiah S, Hoskote M, Ratanawongsa N, Schillinger D. A Randomized Trial to Train Vulnerable Primary Care Patients to Use a Patient Portal. J Am Board Fam Med. 2019 Mar-Apr;32(2):248-258. doi: 10.3122/jabfm.2019.02.180263. PMID 30850461
- [Background] Ramirez V, Johnson E, Gonzalez C, Ramirez V, Rubino B, Rossetti G. Assessing the Use of Mobile Health Technology by Patients: An Observational Study in Primary Care Clinics. JMIR Mhealth Uhealth. 2016 Apr 19;4(2):e41. doi: 10.2196/mhealth.4928. PMID 27095507
- [Background] Schickedanz A, Huang D, Lopez A, Cheung E, Lyles CR, Bodenheimer T, Sarkar U. Access, interest, and attitudes toward electronic communication for health care among patients in the medical safety net. J Gen Intern Med. 2013 Jul;28(7):914-20. doi: 10.1007/s11606-012-2329-5. Epub 2013 Feb 20. PMID 23423453
- [Background] Nishii A, Campos-Castillo C, Anthony D. Disparities in patient portal access by US adults before and during the COVID-19 pandemic. JAMIA Open. 2022 Dec 16;5(4):ooac104. doi: 10.1093/jamiaopen/ooac104. eCollection 2022 Dec. PMID 36540762
- [Background] Barbosa W, Zhou K, Waddell E, Myers T, Dorsey ER. Improving Access to Care: Telemedicine Across Medical Domains. Annu Rev Public Health. 2021 Apr 1;42:463-481. doi: 10.1146/annurev-publhealth-090519-093711. PMID 33798406
- [Background] Meng YY, Diamant A, Jones J, Lin W, Chen X, Wu SH, Pourat N, Roby D, Kominski GF. Racial and Ethnic Disparities in Diabetes Care and Impact of Vendor-Based Disease Management Programs. Diabetes Care. 2016 May;39(5):743-9. doi: 10.2337/dc15-1323. Epub 2016 Mar 10. PMID 26965718
- [Background] Wisniewski H, Gorrindo T, Rauseo-Ricupero N, Hilty D, Torous J. The Role of Digital Navigators in Promoting Clinical Care and Technology Integration into Practice. Digit Biomark. 2020 Nov 26;4(Suppl 1):119-135. doi: 10.1159/000510144. eCollection 2020 Winter. PMID 33442585
- [Background] Samuels-Kalow M, Jaffe T, Zachrison K. Digital disparities: designing telemedicine systems with a health equity aim. Emerg Med J. 2021 Jun;38(6):474-476. doi: 10.1136/emermed-2020-210896. Epub 2021 Mar 4. PMID 33674277
- [Background] Uscher-Pines L, Sousa J, Jones M, Whaley C, Perrone C, McCullough C, Ober AJ. Telehealth Use Among Safety-Net Organizations in California During the COVID-19 Pandemic. JAMA. 2021 Mar 16;325(11):1106-1107. doi: 10.1001/jama.2021.0282. PMID 33528494
- [Background] Jain V, Al Rifai M, Lee MT, Kalra A, Petersen LA, Vaughan EM, Wong ND, Ballantyne CM, Virani SS. Racial and Geographic Disparities in Internet Use in the U.S. Among Patients With Hypertension or Diabetes: Implications for Telehealth in the Era of COVID-19. Diabetes Care. 2021 Jan;44(1):e15-e17. doi: 10.2337/dc20-2016. Epub 2020 Nov 2. No abstract available. PMID 33139408
- [Background] Alkureishi MA, Choo ZY, Rahman A, Ho K, Benning-Shorb J, Lenti G, Velazquez Sanchez I, Zhu M, Shah SD, Lee WW. Digitally Disconnected: Qualitative Study of Patient Perspectives on the Digital Divide and Potential Solutions. JMIR Hum Factors. 2021 Dec 15;8(4):e33364. doi: 10.2196/33364. PMID 34705664
- [Background] Gaskin DJ, Hadley J. Population characteristics of markets of safety-net and non-safety-net hospitals. J Urban Health. 1999 Sep;76(3):351-70. doi: 10.1007/BF02345673. PMID 12607901
- [Background] Khoong EC, Butler BA, Mesina O, Su G, DeFries TB, Nijagal M, Lyles CR. Patient interest in and barriers to telemedicine video visits in a multilingual urban safety-net system. J Am Med Inform Assoc. 2021 Feb 15;28(2):349-353. doi: 10.1093/jamia/ocaa234. PMID 33164063
- [Background] Tieu L, Schillinger D, Sarkar U, Hoskote M, Hahn KJ, Ratanawongsa N, Ralston JD, Lyles CR. Online patient websites for electronic health record access among vulnerable populations: portals to nowhere? J Am Med Inform Assoc. 2017 Apr 1;24(e1):e47-e54. doi: 10.1093/jamia/ocw098. PMID 27402138
- [Background] Tieu L, Sarkar U, Schillinger D, Ralston JD, Ratanawongsa N, Pasick R, Lyles CR. Barriers and Facilitators to Online Portal Use Among Patients and Caregivers in a Safety Net Health Care System: A Qualitative Study. J Med Internet Res. 2015 Dec 3;17(12):e275. doi: 10.2196/jmir.4847. PMID 26681155
- [Derived] Omomukuyo A, Ramirez A, Davis A, Velasquez A, Najmabadi AL, Kong M, Willard-Grace R, Brown W 3rd, Broderick A, Suomala K, McCulloch CE, Franco N, Sarkar U, Lyles C, Tran AS, Sharma AE, Tuot DS. Achieving Chronic Care Equity by Leveraging the Telehealth Ecosystem (ACCTIVATE): A Multilevel Randomized Controlled Trial Protocol. Med Res Arch. 2024 Nov;12(11):6087. doi: 10.18103/mra.v12i11.6087. PMID 39679006